CLINICAL TRIAL: NCT01995591
Title: Prospective Open-label Study Using ex Vivo Injection of ICG to Detect SLN in Patients With Colon Cancer
Brief Title: Indocyanine Green (ICG) in the ex Vivo Detection of Sentinel Lymph Node (SLN)in Colon Cancer
Acronym: 2068
Status: Completed | Type: Observational
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2068
Record Dates: First submitted 2013-11-20; First posted 2013-11-26 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2015-06

CONDITIONS: Colon Cancer; Colon Surgery
Keywords: colon cancer; sentinel lymph node; Indocyanine Green
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Evaluation of the possibility to detect sentinel lymph node(s) after ex vivo Indocyanine Green injections around the tumour in pieces of colectomy from patients with colon cancer.

DETAILED DESCRIPTION:
Primary objective Feasibility study of ex vivo injections of ICG to image and detect the sentinel lymph nodes in patients with colon cancer.

Secondary objectives:

To determine the sensitivity of ICG in the dissected piece of colon cancer compared with the blue dye.

Tertiary objectives:

Evaluation of the influence of this approach on the up-staging of the patients

Microscopic study of the ICG distribution in the lymph nodes (in the lymphatic sinuses, in specific cells, in cancerous foci…)

Methodology:

In the operating room:

Patients will undergo standard surgical resection. Immediately after removal of the colon and node-bearing mesentery, using different 29 Gauge insulin syringes, blue dye (2 ml blue dye: 0.5 ml per injection) and ICG (2 ml with 0,5 mg ICG per ml: 0.5 ml per injection) will be injected in the fresh specimen beside each other submucosally around the tumour in at least four sites (as many injections needed to cover all the perimeter of the tumour) for each agent. The injection sites will be then gently stretched and massaged for 3-5 min to stimulate the tracers to flow along the lymphatic channels. Fluoroscopic imagings of the mesentery will be performed during the injections and during these manoeuvers.

The research and identification of the sentinel lymph nodes will be then performed as follows:

1. he will first localize the blue colored lymph vessels (if visible) as well as the palpable and/or blue colored lymph nodes. These last ones will be marked for dissection with a blue suture.
2. using the PDE camera, he will thereafter localize the fluorescent lymph vessels (if visible) as well as the palpable and/or fluorescent lymph nodes. These last ones will be marked for dissection with a green suture.

Histopathology in the Laboratory of Pathology:

When all SLN are identified, they will be dissected and classified as follows:

* SLN first seen as blue and confirmed also as fluorescent using PDE
* SLN seen as blue but not confirmed to be fluorescent using PDE
* SLN not directly visible as blue but seen fluorescent using PDE (the LN in this group will be controlled for their blue or not character when dissected)
* LN identified by the pathologist as pathological but not blue and not fluorescent.

After the dissection of these SLN, the specimen will be processed as usual using routine procedure for further examination of the non SLN by the pathologists. Once these lymph nodes are dissected, they will be tested for the emitted fluorescence.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histo-pathological diagnosis of colon cancer who are candidate for laparoscopic colectomy,
* Informed consent form signed.

Exclusion Criteria:

* Definite lymph node metastases diagnosed either pre-operatively, or per-operatively
* Inability to give informed consent,
* Age < 18 years old,
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with colon cancer who will have colectomy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-01; Primary Completion 2013-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
number of sentinel lymph nodes identified in pieces of colectomy from patients with colon cancer with Indocyanine Green | 18 monthes

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Liberale, MD, Principal Investigator — Surgeon in Jules Bordet Institute
Locations (1):
- Jules Bordet Institute, Brussels, Brussels Capital, Belgium